CLINICAL TRIAL: NCT01800916
Title: Investigating the Safety and Performance of New 1-piece Ostomy Product Concepts Compared With SenSura 1-piece in Subjects With an Ileostomy
Brief Title: Safety and Performance of New 1-piece Ostomy Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CP236
Record Dates: First submitted 2013-02-22; First posted 2013-02-28 (Estimated); Results first posted 2014-05-30 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Stoma Ileostomy
Keywords: ileostomy; Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment sequence 1 (Experimental): The subjects randomised to Treatment sequence 1 are going to test
  1. Coloplast Adhesive baseplate A (A)
  2. Coloplast Adhesive baseplate B (B)
  3. SenSura 1-piece (S)
  The subjects test the three test products in a randomised order: ABS; BSA; SAB
  Interventions: Device: Coloplast Adhesive baseplate A; Device: Coloplast Adhesive baseplate B; Device: SenSura 1-Piece
- Treatment sequence 2 (Experimental): The subjects randomised to Treatment sequence 2 are going to test
  1. Coloplast Adhesive baseplate B (B)
  2. Coloplast Adhesive baseplate C (C)
  3. SenSura 1-piece (S)
  The subjects test the three test products in a randomised order: CBS; BSC; SCB
  Interventions: Device: Coloplast Adhesive baseplate B; Device: Coloplast Adhesive baseplate C; Device: SenSura 1-Piece
- Treatment sequence 3 (Experimental): The subjects randomised to Treatment sequence 3 are going to test
  1. Coloplast Adhesive baseplate A (A)
  2. Coloplast Adhesive baseplate B (C)
  3. SenSura 1-piece (S)
  The subjects test the three test products in a randomised order: ACS; CSA; SAC
  Interventions: Device: Coloplast Adhesive baseplate A; Device: Coloplast Adhesive baseplate C; Device: SenSura 1-Piece

INTERVENTIONS:
Device: Coloplast Adhesive baseplate A — Coloplast Adhesive baseplate A is a newly developed 1-piece ostomy appliance.
  Arms: Treatment sequence 1; Treatment sequence 3
Device: Coloplast Adhesive baseplate B — Coloplast Adhesive baseplate B is a newly developed 1-piece ostomy appliance
  Arms: Treatment sequence 1; Treatment sequence 2
Device: Coloplast Adhesive baseplate C — Coloplast Adhesive baseplate C is a newly developed 1-piece ostomy appliance
  Arms: Treatment sequence 2; Treatment sequence 3
Device: SenSura 1-Piece — SenSura 1-piece is the commercial CE-marked Coloplast 1-piece SenSura .

SUMMARY:
The aim of the the current investigation is to develop new soft and more flexible 1-piece ostomy products.

DETAILED DESCRIPTION:
The present investigation aims at testing the degree of leakage with the new flexible 1-piece ostomy products as well as other performance and safety parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent and signed letter of authority form.
2. Be at least 18 years of age and have full legal capacity.
3. Be able to handle the bags themselves.
4. Have an ileostomy with a diameter between 15 and 40 mm.
5. Have had their ostomy for at least three months.
6. Currently use a 1-piece flat ostomy appliance with open bag.
7. Use minimum 1 ostomy appliance every second day.
8. Be suitable for participation in the investigation and for using standard adhesive, flat base plate.
9. Must be able to use a custom cut ostomy appliance.
10. Accept to test three 1-piece ostomy appliances in the investigation.
11. Negative result of a pregnancy test for women of childbearing age (only DK).

Exclusion Criteria:

1. Use irrigation during the study (flush the stoma with water).
2. Currently receiving or have within the past 2 months received radio- and/or chemotherapy.
3. Currently receiving or have within the past months received local or systemic steroid treatment in the peristomal area.
4. Are pregnant or breastfeeding.
5. Participating in other interventional clinical investigations or have previously participated in this investigation.
6. Currently using ostomy belt.
7. Currently using extended wear product.
8. Known hypersensitivity towards any of the test products
9. Suffer from peristomal skin problems that preclude participation in the investigation (assessed by the investigation nurse) -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birte Jakobsen, Dr., Principal Investigator — Coloplast A/S
Locations (1):
- Holtedam 3, Humlebæk, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was performed primarily via Coloplast own subject database. In Norway recruitment also took place through medical clinics and hospitals.
Pre-assignment Details: 65 participants were recruited. However, one participant was a screen failure and was not randomized and did not try any products.
Groups:
- Test A/Test B/SenSura: The subjects first tested Coloplast test product A then Coloplast test product B and finally the comparator SenSura
- Test A/Test C/SenSura: The subjects first tested Coloplast test product A then Coloplast test product C and finally the comparator SenSura
- Test B/SenSura/Test A: The subjects first tested Coloplast test product B then SenSura and finally Coloplast test product A
- Test B/SenSura/Test C: The subjects first tested Coloplast test product A then SenSura and finally Coloplast test product B
- Test C/Test B/SenSura: The subjects first tested Coloplast test product C then Coloplast test product A and finally the comparator SenSura
- Test C/SenSura/Test A: The subjects first tested Coloplast test product C then SenSura and finally Coloplast test product A
- SenSura/Test A/Test B: The subjects first tested SenSura then Coloplast test product A and finally Coloplast test product B
- SenSura/Test A/Test C: The subjects first tested SenSura then Coloplast test product A and finally Coloplast test product C
- SenSura/Test C/Test B: The subjects first tested SenSura then Coloplast test product C and finally Coloplast test product B
Period: Test Period 1 (1 Week)
Arm/Group | Test A/Test B/SenSura | Test A/Test C/SenSura | Test B/SenSura/Test A | Test B/SenSura/Test C | Test C/Test B/SenSura | Test C/SenSura/Test A | SenSura/Test A/Test B | SenSura/Test A/Test C | SenSura/Test C/Test B
Started | 7 | 7 | 7 | 7 | 8 | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 6 | 7 | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Convex product user | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Test Period 2 (1 Week)
Arm/Group | Test A/Test B/SenSura | Test A/Test C/SenSura | Test B/SenSura/Test A | Test B/SenSura/Test C | Test C/Test B/SenSura | Test C/SenSura/Test A | SenSura/Test A/Test B | SenSura/Test A/Test C | SenSura/Test C/Test B
Started | 7 | 7 | 7 | 6 | 7 | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 6 | 7 | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Test Period 3 (1 Week)
Arm/Group | Test A/Test B/SenSura | Test A/Test C/SenSura | Test B/SenSura/Test A | Test B/SenSura/Test C | Test C/Test B/SenSura | Test C/SenSura/Test A | SenSura/Test A/Test B | SenSura/Test A/Test C | SenSura/Test C/Test B
Started | 7 | 7 | 7 | 6 | 7 | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 6 | 7 | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data was obtained on the ITT population. Two subjects were not included in the ITT population. One was discovered before randomization (this subject is not found in the Participant flow), the other was randomized before it was seen that the subjects was screen failure and included in the randomized population but not in the ITT population
Arm/Group | Overall Study Population
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Degree of Leakage
Description: The degree of leakage is measured using a 4-point leakage scale developed by Coloplast A/S at every baseplate change.
  The subjects had to tick off one of the following choices:
  1. No leakage
  2. Starting to leak
  3. Leakage
  4. Sudden Leakage
Time Frame: one week
Population: The subjects were randomized to one of nine possible treatment groups. Each group consisted of three equal periods in which the subjects tested two test products and the comparator product (SenSura 1-piece). An equal distribution among the three arms and nine different treatment groups was aimed for. The ITT population was used for the analysis.
Measure: Number; unit: percentage of baseplates with no leakage
Units Other Than Participants: baseplates
Arm/Group | Test A | Test B | Test C | SenSura
Number analyzed (Participants) | 42 | 41 | 42 | 62
Number analyzed (baseplates) | 286 | 280 | 291 | 417
percentage of baseplates with no leakage | 50 | 44 | 41 | 60

ADVERSE EVENTS:
Time Frame: The adverse events were collected during the investigation - up to three weeks
Arm/Group | Test A | Test B | Test C | SenSura
Serious Adverse Events (participants affected / at risk) | 1/42 | 1/42 | 0/42 | 0/62
Other Adverse Events (participants affected / at risk) | 18/42 | 12/42 | 11/42 | 13/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test A (N=42) | Test B (N=42) | Test C (N=42) | SenSura (N=62)
dehydration (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — dehydration due to diarre
obstipation due to parastomal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test A (N=42) | Test B (N=42) | Test C (N=42) | SenSura (N=62)
peristomal skin irritation (Skin and subcutaneous tissue disorders) | 14 (19) | 10 (14) | 7 (8) | 8 (8)
diarre (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
headache (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — not related to product
stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
bleeding from rectum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
otitis left ear (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
gout (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
active colitis ulcerosa in remaining bowl (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
small blister on peristomal skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — not related to product
gastroenterotitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
skin injury on forehead and nose (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — caused by a mountain bike accident
pertussis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less